CLINICAL TRIAL: NCT04865926
Title: Comparison Of The Neck And Scapular Proprioceptive Neuromuscular Facilitation Exercises On Postural Disorders, Scapular Dyskinesia And Round Shoulders in Individuals With Cervical Sagittal Alignment Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0287
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Forward Head Posture; Sagittal Cervical Malalignment; Rounded Shouler; Scapular Dyskinesis
Keywords: Forward head posture; Proprioceptive Neuromuscular Facilitation; Mckenzie; Kendall

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular and Neck Proprioceptive Neuromuscular Facilitation Group (Experimental): Participants in the intervention group will be applied neck and scapular Proprioceptive Neuromuscular Facilitation exercises lasting 40 minutes for 3 sessions a week for 4 weeks.
  Interventions: Other: Scapular and Neck Proprioceptive Neuromuscular Facilitation exercises
- Control Group (Experimental): McKenzie and Kendall exercises will be given to the participants in the control group. Exercises will be done 3 sessions a week over a 4-week period.
  Interventions: Other: McKenzie and Kendall exercises

INTERVENTIONS:
Other: Scapular and Neck Proprioceptive Neuromuscular Facilitation exercises — The researcher will perform a total of 12 sessions of scapular and neck pnf exercises for 4 weeks. The participants will apply PNF exercises using rhythmic initiation, rhythmic stabilization and cobination techniques of isotonics. Patterns of anterior elevation, posterior depression, anterior depression, posterior elevation will be used in scapular exercises. Upper cervical flexion, lower cervical flexion, rotation and lateral flexion patterns will be used in neck pnf exercises.
  Arms: Scapular and Neck Proprioceptive Neuromuscular Facilitation Group
Other: McKenzie and Kendall exercises — Kendall and Mckenzie exercises will be given to the participants as a home workout. The self-stretch exercise methods are as followed: Placing both hands on the shoulders and pushing out the chest, placing one hand over the shoulder and grasp the elbow of the turned hand, with the other hand over the head and slowly pull it inward, throwback the head until it has reached the fully stretched point, look straight ahead and slowly turn the head horizontally until the maximum value is reached, throwback the head, and turn it until it has reached the fully stretched point, lower the head turn it until it has reached the maximal point. Stretching pectoralis muscle, strengthening shoulder retraction, strengthening the deep cervical flexors, strengthening the deep cervical flexors.
  Arms: Control Group

SUMMARY:
In modern society, repetitive and monotonous activities are increasing due to the decrease in general physical activity, the development of the information technology industry, and time culture flow. Therefore, prolonged exposure to unstable or abnormal posture can trigger a chain reaction of poor alignment and imbalance, leading to musculoskeletal diseases such as muscle stiffness or repetitive traumatic injury.

Sagittal cervical malalignment (SCM), and also known as Forward head posture (FHP), is one of the poor posture types of the head commonly seen in the sagittal plane. İt is defined as the forward shift of the head. As the head moves forward, the center of gravity changes. To compensate for this shift in the center of gravity, the upper body slides back and the shoulders move forward, the rounded shoulder develops so that the head is placed in front of the body.

SCM can cause many harmful symptoms such as neck pain, shoulder pain, back pain, chronic headaches, increased curvature of the spine and scapular dyskinesis, and rounded shoulder.

DETAILED DESCRIPTION:
Proper posture is defined as musculoskeletal balance with minimal stress or strain on the body. The human body is a multi-joint system with kinetic chains controlled by the central nervous system, with a series of joints that interact with muscle activity.

Prolonged exposure to unstable or abnormal posture can trigger a chain reaction of weak alignment and imbalance, leading to musculoskeletal diseases such as muscle stiffness or repeated traumatic injury. Sagittal cervical malalignment (SCM), in other words forward head posture (FHP), is one of the poor posture types of the head commonly seen in the sagittal plane. It is defined as the shift of the center of the head towards the front. As the head moves forward, the center of gravity changes. To compensate for this shift in the center of gravity, the upper body slides back and the shoulders move forward, the rounded shoulder develops so that the head is placed in front of the body.

SCM of the head is defined as the anterior extension of the head with hyperextension of the upper cervical vertebrae (C1-C3) and flexion of the lower cervical vertebrae (C4-C7) and hyperlordosis of the cervical curve. It can be caused by a variety of factors, including Sleeping in positions with an excessive elevation of the head, prolonged use of the computer, and developed back muscle weakness.

SCM can cause many harmful symptoms such as neck pain, shoulder pain, back pain, chronic headaches, increased curvature of the spine and scapular dyskinesia, and rounded shoulder.

The rounded shoulder is a bent posture in which the scapulae are elevated and the acromion protrudes forward compared to the center of gravity of the body. These changes can cause an imbalance of the surrounding muscles and eventually pain in the head, temporomandibular joints, neck, back, shoulders and arms.

Scapular dyskinesia is referred to as visible changes in scapular position and movement patterns. It produces changes in the kinematics of the glenohumeral and acromioclavicular joints and can interfere with the activity of the periscapular muscles and rotator cuffs.7 Proprioceptive neuromuscular facilitation (PNF) methods focus on functional diagonal movement patterns and use cutaneous, visual, and auditory stimulation to improve neuromuscular control and function as well as muscle strength, balance, and flexibility. It is used as a progressive resistance for functional training in therapeutic exercises, improves joint limitations, and strengthens muscles. Scapular and neck PNF patterns are known to increase the stability of the head, neck, and scapular muscles.

ELIGIBILITY:
Inclusion Criteria:

* Those with a Kraviovertebral angle below 50o.
* Healthy individuals who have not had an upper extremity injury in the last 6 months.
* Has 3 or more pain in VAS for at least 3 months

Exclusion Criteria:

* Have received any physiotherapy program in the last 6 months due to neck pain or back pain.
* With structural scoliosis
* Have a history of fracture in the cervical vertebrae
* Have any rheumatic disease affecting the neck
* Having had a cervical spine surgery
* Spinal cord compression from a tumor or other cause
* Those with neurological deficits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angel Evaluation | 5 minutes
  The anatomical points of the participant's ipsilateral tragus and C7 spinous process will be marked. The angle between the line connecting the C7 spinous process and the tragus point and the horizontal line drawn from C7 gives the craniovertebral angle. Individuals with a CVA angle of less than 50 degrees are individuals with cervical sagittal alignment. A camera will be placed at a distance of 1 meter and the camera lens will be at the C7 level, fınally the lateral photos of the patients will be taken. Angle calculations will be made using the triangular screen ruler computer program of Markus Bader- MB Software Solutions.

SECONDARY OUTCOMES:
Neck Pain assessment | 1 minute
  Neck pain intensity will be objectively evaluated with the Visual Analogue Scale. The patient will be asked to mark the severity of the pain felt on the line drawn with a 10 cm ruler such as 0 = "no pain" 10 = "very severe pain".
The International Physical Activity Questionnaire (IPAQ)- Short Form | 3 minutes
  This short-form consists of 7 questions and provides information about sitting, walking, moderately vigorous activities, and time spent on vigorous activities. In the IPAQ short form evaluation, the energy required for the activities will be calculated with the MET-minute score.
Neck disailty index (NDİ) | 3 minutes
  It is a questionnaire consisting of 10 topics investigating how neck pain affects the daily life of the patient. These headings evaluate the severity of pain, personal care, carrying, reading, headache, concentration, work-life, driving, sleep and recreation. Each section is scored between 0 and 5. The total score of NDİ is calculated over 100. According to the BDI score; 0-8% no disability, 10-28% mild disability, 30-48% moderate disability, 50% 68 severe disability, 68% over full disability.
Active Cervical Range of Motion | 10 minutes
  Active cervical range of motion is measured with goniometer application (G-pro© ), which was proven to be valid by Pourahmadi in 2018. For measuring flexion and extension, the testing position of the iPhone was placed just beside the external auditory meatus, and one axis of the app was aligned with the imaginary line between the base of the nostril and the external auditory meatus. Active lateral flexion range of motion was measured in the sitting position. The center of the app was placed over the C7 spinous process and one axis of the app was aligned with the occipital protuberance. Finally, active craniocervical rotation in sitting, this movement was evaluated in the supine position the center of the app was positioned at the center of the head and one axis was aligned with the nose.
Evaluation of Postural Problems | 5 minutes
  In the study, the photography method will be used in measuring the tilt angle, the frontal tilt angle of the head, and the rounded shoulder angle. The determined anatomical points will be marked, the lateral and anterior photographs of the patients will be taken with a digital camera. Angular calculations will be made using the triangular screen ruler computer program of Markuz Bader- MB Software Solutions.
  Head tilt, will be calculated by finding the angle between the line drawn between the endpoint of the eye from the tragus point and the horizontal line drawn from the tragus line.
  Frontal tilt angle is the angle formed between the line joining the lower edges of each ear and the horizontal line Rounded shoulder, is calculated by finding the angle between the line joining the C7 spinous process and the acromion midpoint, and the horizontal line drawn from the midpoint of C7.
Lateral Scapular Slide Test | 10 minutes
  Each subject was instructed to actively achieve the first test position both arms at the sides in glenohumeral joint neutral, second position subject actively placed both hands on the ipsilateral hips and place the humerus in medial rotation at 45° of abduction in the coronal plane and third position subject actively extended both elbows, placed the upper extremities in a position of maximum medial rotation at 90° of abduction in the coronal plane. When the test position will be obtained the inferior angle of the scapula and the adjacent spinous process of the reference vertebra in the same horizontal plane will be identified through palpation and measured with a digital caliper bilaterally.
The Craniocervical Flexion Test | 10 minutes
  The test is performed with the patient in supine crook lying with the neck in a neutral position such that the line of the face is horizontal and a line bisecting the neck longitudinally is horizontal to the testing surface. The uninflated pressure sensor is placed behind the neck so that it abuts the occiput and is inflated to a stable baseline pressure of 20 mm Hg, a standard pressure sufficient to fill the space between the testing surface and the neck but not push the neck into a lordosis. The device provides feedback and direction to the patient to perform the required five stages of the test. The patient is instructed that the test is not one of strength but rather one of precision. The movement is performed gently and slowly as a head-nodding action (as if saying "yes").

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus